CLINICAL TRIAL: NCT02144779
Title: Improving Family Outcomes With a Communication Intervention in the Pediatric ICU
Brief Title: Family Communication and Support in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ross Hays (Other)
Responsible Party: Sponsor-Investigator, Ross Hays, MD, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1RO1NRO11179
Record Dates: First submitted 2014-05-14; First posted 2014-05-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Reducing Post Traumatic Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): No treatment for this group
  Interventions: Behavioral: Usual Care
- Assigned to palliative care team (Experimental): The intervention group will be assigned to a palliative care team member that will facilitate communication and meetings between families and the medical team
  Interventions: Behavioral: Assigned to palliative care team

INTERVENTIONS:
Behavioral: Assigned to palliative care team — Communication and Support through the palliative care team assigned to intervention participants.
  Arms: Assigned to palliative care team
Behavioral: Usual Care — usual hospital care, not assigned to palliative care team
  Arms: Usual care

SUMMARY:
This project is evaluating the effect of a standardized communication intervention in the pediatric intensive care unit (PICU) on long-term distress of family members of children in the PICU for 5 days or longer. The study hypothesis is that intervention families will have lower (better) acute stress disorder scores when their child is discharged from the PICU and lower (better) post-traumatic stress disorder scores at 3-month follow-up, as compared to the control group families. The investigators will recruit 220 families (110 in each of the control and intervention groups). Families who are randomized to the intervention group will receive routine visits from members of the PACT (palliative care) team at least three times/week to address psychosocial needs, keep families informed about their child's health status, and offer emotional and instrumental support and resources. Families in the control group will receive usual care in the PICU. The intervention will end whenever the child is discharged from the PICU, which usually happens within 3 weeks of enrollment. The investigators will assess family outcomes at discharge from the PICU and 90 days after study enrollment. The investigators will conduct two additional activities to learn more about the processes of care for those in both the intervention and control groups. First, during the intervention, the investigators will recruit 30 families (15 in each group) and ask permission to audio-record the family care conferences to assess communication styles and gain greater insight into the differences in practice with or without the participation of the intervention team. The investigators will obtain additional consent from participants in these family conferences who are not otherwise enrolled in the study. Second, after completion of the 3-month follow-up interview, a sub-sample of a different 30 families (again, 15 in each group) will be invited to participate in qualitative interviews to debrief about their experience in the study and the intervention (for those in that group). This will be a one-time interview scheduled within 60 days of recruitment for this part of the project.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* actively involved in the life of the patient receiving care; and
* functionally fluent in English or Spanish.

Exclusion Criteria:

* discharge plan in place for patient before day 4
* previously received palliative care
* patient placed on extracorporeal membrane oxygenation (ECMO)
* no prior admission to ICU for same hospitalization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder | 90 days after baseline
  PTSD will be measures using the Post Traumatic Stress Disorder (PCL-C) scale.

SECONDARY OUTCOMES:
Acute Stress Disorder | Baseline, and up to 90 days after
  Will be measured using the Acute Stress Disorder Scale
Communication Satisfaction | Baseline, and up to 90 days after
  Questions will be asked about family satisfaction with provider communication.
Conflict | Baseline and up to 90 days after
  Questions will be asked about conflict with providers.

OTHER OUTCOMES:
Mental Health Symptoms | Baseline and up to 90 days after
  Will be measured with the PHQ-9 (Depression) and GAD-7 (Anxiety) scales.
Family Relationship | Baseline and up to 90 days after
  Will be measured using the Family relationship index
Social Support | Baseline and up to 90 days after
  Will be measured using the Perceived Social Support scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hays, MD, Principal Investigator — Seattle Childrens Hospital
Locations (1):
- Seattle Childrens Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Doorenbos A, Lindhorst T, Starks H, Aisenberg E, Curtis JR, Hays R. Palliative care in the pediatric ICU: challenges and opportunities for family-centered practice. J Soc Work End Life Palliat Care. 2012;8(4):297-315. doi: 10.1080/15524256.2012.732461. PMID 23194167
- [Background] Doorenbos AZ, Starks H, Bourget E, McMullan DM, Lewis-Newby M, Rue TC, Lindhorst T, Aisenberg E, Oman N, Curtis JR, Hays R; Seattle Ethics in ECLS (SEE) Consortium; Clark JD, Baden HP, Brogan TV, Di Gennaro JL, Mazor R, Roberts JS, Turnbull J, Wilfond BS. Examining palliative care team involvement in automatic consultations for children on extracorporeal life support in the pediatric intensive care unit. J Palliat Med. 2013 May;16(5):492-5. doi: 10.1089/jpm.2012.0536. Epub 2013 Mar 29. PMID 23540309
- [Derived] Iwata M, Han S, Hays R, Doorenbos AZ. Predictors of Depression and Anxiety in Family Members 3 Months After Child's Admission to a Pediatric ICU. Am J Hosp Palliat Care. 2019 Oct;36(10):841-850. doi: 10.1177/1049909119859517. Epub 2019 Jun 30. PMID 31256606
- [Derived] Starks H, Doorenbos A, Lindhorst T, Bourget E, Aisenberg E, Oman N, Rue T, Curtis JR, Hays R. The Family Communication Study: A randomized trial of prospective pediatric palliative care consultation, study methodology and perceptions of participation burden. Contemp Clin Trials. 2016 Jul;49:15-20. doi: 10.1016/j.cct.2016.05.004. Epub 2016 Jun 1. PMID 27263074